CLINICAL TRIAL: NCT02600260
Title: Thromboprophylaxis in Pregnant Women in Hospital: A Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, VENINA ISABEL POÇO VIANA LEME DE BARROS, MD, PhD, Group of Thrombosis and Thrombophilia in pregnancy, Clinics Hospital, University of Sao Paulo, University of Sao Paulo General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 37431414.9.0000.0068
Record Dates: First submitted 2015-10-30; First posted 2015-11-09 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Thrombophilia Associated With Pregnancy; Perioperative/Postoperative Complications; Venous Thrombosis; Pulmonary Embolism; Other Specified Risk Factors in Pregnancy; Deep Vein Thrombosis
Keywords: thrombophilia; thrombosis; Pregnancy, High-Risk; venous thrombosis; enoxaparin; risk assessment; deep vein thrombosis; pulmonary embolism; hospitalization
MeSH Terms: conditions — Postoperative Complications; Venous Thrombosis; Pulmonary Embolism; Thrombophilia; Thrombosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- enoxaparin (Other): A prospective study that will evaluate all pregnant women admitted for clinical treatment and / or surgery through the application of a thromboprophylaxis protocol with risk assessment score.The patient in whom prophylaxis would be indicated are those with scores greater than or equal to 3. The drug to be used is enoxaparin and the dose to be used depends on the weight of the patient.It will be further assessed: adverse effects of treatment with enoxaparin, protocol failure in the group treated and untreated (without anticoagulation) and bleeding incidence in both groups.
  Interventions: Drug: Enoxaparin
- no intervention (Other): Pregnant women admitted in hospital for clinical treatment and/or delivery and that does not score for thromboprophylaxis.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Enoxaparin — Patients who score higher or equal to 3, receive a prophylactic dose of enoxaparin. The first dose of enoxaparin is administered 8 hours after vaginal or abdominal delivery. Subsequent doses are administered daily for up to 15 days. The dose depends on patient weight.
  Other Names: lovenox; clexane
  Arms: enoxaparin
Other: No intervention — Hospitalized patients that score less than three are not prescribed enoxaparin.
  Other Names: No enoxaparin; Score lower than three
  Arms: no intervention

SUMMARY:
Hospitalization in pregnancy and childbirth greatly increases the thromboembolic risk of these patients. The application of a protocol for assessing the risk of VTE reduces mortality and morbidity of these phenomena.

DETAILED DESCRIPTION:
Thromboembolic events are among the leading causes of maternal morbidity and mortality in pregnancy / postpartum period. They are the leading cause of maternal death in developed countries. Risk factors for venous thromboembolism (VTE) during pregnancy and postpartum as family history or personal history of VTE, thrombophilia, age over 35, obesity and high parity has been the most studied. One of the main risk factors is hospitalization, which increases up to 20 times the risk of VTE.

Objective: The objective of the study is to identify early risk factors for VTE in hospitalized pregnant women and institute appropriate prophylaxis to reduce the incidence and morbidity.

Methods: A prospective study that will evaluate all pregnant women admitted for clinical treatment and / or surgery in the Department of Obstetrics and Gynecology, Clinics Hospital, University of São Paulo through the application of a thromboprophylaxis protocol with risk assessment score. The patient in whom prophylaxis would be indicated are those with scores greater than or equal to 3. The drug to be used is enoxaparin and the dose to be used depends on the weight of the patient.

It will be further assessed: adverse effects of treatment with enoxaparin, protocol failure in the group treated and untreated (without anticoagulation) and bleeding incidence in the untreated group.

Risk score description: score 3 - previous thrombosis/thromboembolism, homozygous mutations, combined thrombophilia risk factors, antiphospholipid syndrome, cancer(stomach, pancreas, lung), inflammatory conditions, lupus, sickle cell disease, nephrotic syndrome, heart disease; Score 2 - Protein C deficiency, Protein S deficiency, heterozygous F5 Leiden, heterozygous F2 G20210A mutation, cancer(last 6 months), chemotherapy(last 6m), immobility, bed rest >4d prior to C-section, current serious infections, BMI≥40 kg/m2 , age≥40y, lung disease(cyanosis), postpartum hemorrhage >1L; Score 1 - age ≥ 35 and ≤39 y, parity ≥3, multiple pregnancy, hyperemesis, gross varicose veins, smoker ≥20, surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant women hospitalized.

Exclusion Criteria:

* Previous use of anticoagulation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7212 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Number of hospitalized pregnant patients with venous thromboembolism (VTE), death and adverse events after applying an in hospital risk score for thrombosis at 12 weeks post discharge. | 4 years
  Identify early risk factors for VTE in hospitalized pregnant women and prescribe appropriate prophylaxis to reduce the incidence, morbidity and mortality of VTE. The patients that score ≥ 3 will receive enoxaparin. This group will be analyzed for the incidence of adverse outcomes: VTE, bleeding, death until 3 months post hospitalization. This same analysis will be done in those patients who have not received heparin. The patients that could not receive heparin due to bleeding risk will be analyzed also. The analysis of the score will also describe if the higher the score, the higher the index of adverse events, mainly when it is not possible to prescribe the prophylaxis.

CONTACTS AND LOCATIONS:
Overall Officials: Venina V Barros, MD, PhD, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- University of Sao Paulo General Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Royal College of Obstetricians and Gynaecologists. Reducing the risk of thrombosis and embolism during pregnancy and the puerperium. Green-top Guideline No. 37a 2009.
- [Background] Bates SM, Greer IA, Middeldorp S, Veenstra DL, Prabulos AM, Vandvik PO. VTE, thrombophilia, antithrombotic therapy, and pregnancy: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e691S-e736S. doi: 10.1378/chest.11-2300. PMID 22315276
- [Background] Abbasi N, Balayla J, Laporta DP, Kezouh A, Abenhaim HA. Trends, risk factors and mortality among women with venous thromboembolism during labour and delivery: a population-based study of 8 million births. Arch Gynecol Obstet. 2014 Feb;289(2):275-84. doi: 10.1007/s00404-013-2923-8. Epub 2013 Jul 18. PMID 23864199
- [Result] Hase EA, Barros VIPVL, Igai AMK, Francisco RPV, Zugaib M. Risk assessment of venous thromboembolism and thromboprophylaxis in pregnant women hospitalized with cancer: Preliminary results from a risk score. Clinics (Sao Paulo). 2018 Oct 18;73:e368. doi: 10.6061/clinics/2018/e368. PMID 30365820
- [Result] Barros V, Igai A, Fernanda B, Bortolotto M, Francisco R, Zugaib M. Preventing Maternal Death and Morbidity from Venous Thromboembolism (VTE): Results from a VTE Risk Score Trial during Hospitalization [abstract]. Res Pract Thromb Haemost. 2020; 4 (Suppl 1). https://abstracts.isth.org/abstract/preventing-maternal-death-and-morbidity-from-venous- thromboembolism-vte-results-from-a-vte-risk-score-trial-during-hospitalization/. Accessed August 6, 2020.